CLINICAL TRIAL: NCT00987727
Title: Safety and Efficacy of Carboxymethylcellulose for Ocular Surface Integrity in Symptomatic Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Vice President Medical Affairs, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAF-AGN-OPH-DE-011
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-08

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Carboxymethylcellulose Sodium; Glycerol; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): carboxymethylcellulose 0.5% and glycerin 0.9% (OPTIVE® MD)
  Interventions: Drug: carboxymethylcellulose 0.5% , glycerin 0.9% (OPTIVE® MD)
- 2 (Active Comparator): sodium hyaluronate 0.18% (VISMED® Multi)
  Interventions: Drug: sodium hyaluronate 0.18% (VISMED® Multi)

INTERVENTIONS:
Drug: carboxymethylcellulose 0.5% , glycerin 0.9% (OPTIVE® MD) — One drop in each eye three to six times daily, as needed
  Other Names: OPTIVE® MD
  Arms: 1
Drug: sodium hyaluronate 0.18% (VISMED® Multi) — One drop in each eye three to six times daily, as needed
  Other Names: VISMED® Multi
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of OPTIVE® MD for ocular surface integrity in symptomatic dry eye condition in absence of obvious eye-lid inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Have been using artificial tears for at least 3 months prior to study inclusion
* Have been using preservative free artificial tears at least three times daily (TIB) for at least 2 weeks immediately prior to study inclusion
* Having moderate to severe symptoms suggestive of dry eye

Exclusion Criteria:

* Current enrollment in an investigational drug or device study or participation in such a study within 3 months prior to entry into this study
* Moderate to severe blepharitis
* History or active signs of ocular trauma, ocular infection, or ocular inflammation within the last 3 months
* History or active signs of ocular allergic disease or ocular herpes within the last year
* History or active signs of severe or serious ocular conditions such as inflammatory corneal ulcers, recurrent erosions, and uveitis at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD): carboxymethylcellulose 0.5% and glycerin 0.9% (OPTIVE® MD)
- Sodium Hyaluronate 0.18% (VISMED® Multi): sodium hyaluronate 0.18% (VISMED® Multi)
Period: Overall Study
Arm/Group | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) | Sodium Hyaluronate 0.18% (VISMED® Multi)
Started | 41 | 41
Completed | 36 | 34
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) | Sodium Hyaluronate 0.18% (VISMED® Multi) | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Customized [Number; unit: participants]
  <65 years | 22 | 29 | 51
  >=65 years | 19 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Global Ocular Staining Score at Day 35
Description: Change from baseline in global ocular staining score (range from 0-15) at Day 35. The global ocular staining score is the sum of three different staining severities, each with a score of 0-5 on a 6-point scale, where 0 is no staining (best) and 5 is diffuse staining (worst).
Time Frame: Baseline, Day 35
Population: Per Protocol: All subjects who were randomised, who received at least one dose of the study product, had at least one follow-up visit and who did not have significant protocol violations and who completed the assessment of this outcome measure at Day 35.
Measure: Mean (Standard Deviation); unit: Number on a scale (score)
Arm/Group | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) | Sodium Hyaluronate 0.18% (VISMED® Multi)
Number analyzed (Participants) | 37 | 29
Number on a scale (score)
  Baseline | 5.4 (1.59) | 5.9 (1.47)
  Day 35 | -1.8 (1.95) | -1.8 (2.30)

2. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Questionnaire Score at Day 35
Description: Change from baseline in Ocular Surface Disease Index (OSDI) questionnaire score at Day 35. The OSDI questionnaire consists of 12 questions measuring the presence of ocular symptoms. Each of the 12 questions is assessed using a 5-point scale (where 0=none of the time and 4=all of the time). The score is converted to a 0-100 point score where 0 is no symptoms and 100 is most symptoms.
Time Frame: Baseline, Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number on a scale (score)
Arm/Group | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) | Sodium Hyaluronate 0.18% (VISMED® Multi)
Number analyzed (Participants) | 37 | 27
Number on a scale (score)
  Baseline | 49.05 (17.060) | 51.98 (18.164)
  Day 35 | -13.58 (19.047) | -13.66 (16.542)

ADVERSE EVENTS:
Description: The safety population included all subjects who were randomized and treated with at least one dose of the study product. (Note: 3 randomized subjects in the VISMED® Multi group did not receive a dose and were not included in the safety population).
Arm/Group | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) | Sodium Hyaluronate 0.18% (VISMED® Multi)
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/38
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose 0.5% and Glycerin 0.9% (OPTIVE® MD) (N=41) | Sodium Hyaluronate 0.18% (VISMED® Multi) (N=38)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo